CLINICAL TRIAL: NCT01565681
Title: A Phase 1 Single Ascending Dose Study of ASKP1240 in Healthy Male and Female Volunteers
Brief Title: Study of ASKP1240 After a Single Intravenous Dose at Escalating Dose Levels in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 7163-CL-0101
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Pharmacokinetics of ASKP1240; Healthy Volunteers
Keywords: Healthy Volunteers; B cell CD40 receptor occupancy; anti-CD40 monoclonal antibody
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (13):
- Arm A: ASKP1240 lowest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm B: ASKP1240 second lowest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm C: ASKP1240 third lowest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm D: ASKP1240 fourth lowest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm E: ASKP1240 fifth lowest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm F: ASKP1240 middle dose (Experimental)
  Interventions: Drug: ASP1240
- Arm G: ASKP1240 sixth highest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm H: ASKP1240 fifth highest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm I: ASKP1240 fourth highest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm J: ASKP1240 third highest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm K: ASKP1240 second highest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm L: ASKP1240 highest dose (Experimental)
  Interventions: Drug: ASP1240
- Arm M: Placebo (Placebo Comparator): Sodium Chloride solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1240 — infusion
  Arms: Arm A: ASKP1240 lowest dose; Arm B: ASKP1240 second lowest dose; Arm C: ASKP1240 third lowest dose; Arm D: ASKP1240 fourth lowest dose; Arm E: ASKP1240 fifth lowest dose; Arm F: ASKP1240 middle dose; Arm G: ASKP1240 sixth highest dose; Arm H: ASKP1240 fifth highest dose; Arm I: ASKP1240 fourth highest dose; Arm J: ASKP1240 third highest dose; Arm K: ASKP1240 second highest dose; Arm L: ASKP1240 highest dose
Drug: Placebo — infusion
  Other Names: Sodium Chloride solution
  Arms: Arm M: Placebo

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of ASKP1240 after a single intravenous dose at escalating dose levels in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject weighs at least 50 kg, and has a body mass index (BMI) of 18 to 32 kg/m2 inclusive
* The female subject must be of non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year with follicle stimulating hormone [FSH] > 40 U/L)
* Male subject agrees to no sperm donation until end of study or 90 days post dose, whichever is longer
* The subject is highly likely to comply with the protocol and complete the study
* The subject has a negative urine screen for drugs of abuse, and negative blood or breathalyzer alcohol screen at Screening and clinic admission on Day 1

Exclusion Criteria:

* The subject has a history of severe allergic or anaphylactic reactions
* The subject has history of consuming more than 14 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits)
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check in
* The subject has a supine mean systolic blood pressure < 90 or > 160 mmHg and a mean diastolic blood pressure < 50 or > 90 mmHg, or pulse rate higher than 100 beats per min (bpm), either at screening or clinic check in (blood pressure measurements taken in triplicate after subject has been resting in a supine position for a minimum of 5 minutes)
* The subject is known positive for human immunodeficiency virus (HIV) antibody
* The subject has a positive test for hepatitis C antibody, or for hepatitis B virus surface antigen (HBsAg)
* The subject has at screening or clinic check in that:

  1. white blood cell count (WBC) is < 3.5 or > upper limit of normal
  2. absolute neutrophil count (ANC) is <1.5 or > upper limit of normal
  3. platelet count (PLT) is outside the normal limit
  4. serum creatinine, total bilirubin, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) are > upper limit of normal
  5. creatine phosphokinase (CPK) is > two times upper limit of normal
  6. international normalized ratio (INR) is > upper limit of normal
  7. OR remaining laboratory tests are outside the normal limits and considered by the investigator to be clinically significant with regard to the remaining per protocol laboratory tests
* The subject has received a vaccine within 60 days prior to study drug administration
* The subject has received any systemic immunosuppressant agent within 6 months prior to study drug administration.
* The subject has received any antibody or biologic product within 6 months prior to study drug administration
* The subject has received any systemic steroid within 2 months prior to study drug administration
* The subject has had treatment with prescription or non-prescription drugs, including complementary and alternative medicines (CAM) and excluding over-the-counter (OTC) allergy medications, nasal steroids, nasal inhalers, oral contraceptives, stable hormone replacement therapy (HRT; per Investigator judgment and dose change not expected during study), and intermittent acetaminophen, within 14 days prior to study drug administration
* The subject has received an experimental agent within 30 days or ten half-lives, whichever is longer, prior to study drug administration
* The subject is participating in another clinical trial or has participated in another dose group of the current trial
* The subject has donated or has had significant blood loss or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to dosing
* The subject has a history of heavy smoking or has used tobacco-containing products and nicotine or nicotine-containing products in the past six months prior to Screening
* The subject has a history of thromboembolic or vascular disease especially deep vein thrombosis, pulmonary embolism and varices
* The subject has a positive test for tuberculosis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic variable: Individual subject cell surface antigen (CD40) occupancy levels over time | Days 1-3, 5, 8,15, 22, 29, 43, 60, 75, and 90
  binding of ASKP1240-biotin to B cells
Pharmacokinetics profile: AUCinf and Cmax | Days 1-8,15, 22, 29, 43 and 60
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUCinf) and Maximum concentration of study drug (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetics profile: AUClast, tmax, t1/2, Vz, and CLtot | Days 1-8,15, 22, 29, 43 and 60
  Area under the plasma concentration-time curve from time 0 up to the last quantifiable concentration (AUClast),Time to attain Cmax (tmax), Apparent terminal elimination of half-life (t1/2), Apparent volume of distribution ( Vz), and Total body clearance (CLtot)
Total lymphocyte count | Day -1, Days 1-3, 5, 8,15, 22, 29, 43, and 60
  product of the white blood count (WBC) and percent lymphocytes [from differential]
Peripheral lymphocyte subset quantification | Day -1, Days 1-3, 5, 8,15, 22, 29, 43, and 60
  leukocycte phenotypes: CD3, CD4, CD8,CD16, and CD20
Safety assessed by recording adverse events, laboratory assessments, vital signs, electrocardiograms (ECGs), physical examination, pulse oximetry, and incidence of anti-ASKP1240 antibody formation | Up to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel, Baltimore, Maryland, United States